CLINICAL TRIAL: NCT00718705
Title: Reduction of Spontaneous Prematurity: Impact of Antibiotic Treatment (Josamycin) in Case of Positive PCR for Ureaplasma Spp and/or Mycoplasma Hominis in Amniotic Fluid
Brief Title: Reduction of Spontaneous Prematurity by Antibiotic Treatment (Josamycin)
Acronym: PREMYC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P060216
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-05

CONDITIONS: Prematurity
Keywords: Prematurity; Ureaplasma spp; Mycoplasma Hominis; Amniotic fluid; Josamycine
MeSH Terms: conditions — Premature Birth | interventions — Josamycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): josamycin
  Interventions: Drug: Josamycin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Josamycin — josamycin with posology of 2 grams per day by oral way during 10 days
  Arms: 1
Drug: Placebo — Placebo with posology of 2 grams per day by oral way during 10 days
  Arms: 2

SUMMARY:
The purpose of this study is to test the effectiveness of an antibiotic treatment (Josamycin) in the case of positive PCR for Ureaplasma spp. and/or Mycoplasma hominis in the second quarter on the risk of premature birth.

DETAILED DESCRIPTION:
Infection would be the cause of 40 % of spontaneous premature deliveries. The physiopathological hypothesis accepted is a premature ascent of present bacteria in the low genital ways towards the decidual, the foetal membranes then the amniotic liquid. These bacteria are responsible for an inflammatory reaction to the interface feto-maternal characterized by the production of proinflammatory cytokines and pro-contractants agents (prostaglandins, oxytocin) by the decidual and the membranes.

These mediators cause uterine contractions, a maturation of the uterine collar, a rupture of the membranes then a premature birth.

Several recent publications show on the one hand that Mycoplasma hominis and Ureaplasma spp. are the bacteria most frequently found in the amniotic liquid in the second quarter of the pregnancy and that a positive PCR for these bacteria is associated with a premature birth.

A probable assumption would be that Mycoplasma hominis or Ureaplasma spp. cause a premature birth by infecting the fetal membranes and the decidual, then activating the immune system and the pro-inflammatory production of cytokines. These bacteria are sensitive to antibiotic treatment.

Nevertheless, no randomized controlled trials have been carried out to determine wether an antibiotic treatment would decrease spontaneous prematurity in the case of positive PCR in the amniotic liquid.

ELIGIBILITY:
Inclusion Criteria:

* Patient older ≥ 18 years
* French speaking
* Women who have an amniocentesis between 15 and 20 weeks of amenorrhoea for an antenatal diagnosis
* Affiliated to social security or an equivalent system
* Karyotype analysis and ultrasound morphological normal (apart from minor signs of trisomy 21)
* Clear amniotic fluid (not contaminated by the mother's blood)
* Gestational age is between 15 WA(day+0) and 20 WA(day+6)
* Patient have not allergy to macrolides
* Do not have cure underway by macrolide
* Patient followed during her pregnancy in an investigator site
* Informed consent and signed

Exclusion Criteria:

* No speaking french
* Having an allergy to macrolides
* Having a multiple pregnancy
* Morphological Anomaly
* Patient no consented
* Lactose Intolerance
* Not agreed to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Premature birth | between 22 and 37 completed weeks of pregnancy.

SECONDARY OUTCOMES:
Antenatal :occurence of a miscarriage late | between 16 and 22 weeks of amenorrhoea
Antenatal : premature delivery | at week of amenorrhea <= 34, 32, 28
Antenatal : hospitalisation for risk of premature delivery | antenatal period
antenatal : Number of day of hospitalisation for risk of premature delivery | antenatal period
Antenatal : premature rupture of membranes | before 37 week of amenorrhea
Antenatal : occurence of chorioamnionitis defined by 2 of the following criteria :maternal temperature > 38°C, uterine contractions, Fetid leucorrhoeas, foetal tachycardia > 160bpm, C reactive protein >10mg/l | antenatal period
During childbirth : Hyperthermia > 38°C | Childbirth period
During childbirth : fetal tachycardia > 160 bpm | childbirth period
Post-partum : Hyperthermia > 38°C for more than 24hours | post partum period
Post partum :need an antibiotic treatment for more than 48 hours | post partum period
Neonatal : neonatal mortality late | from day 7 to day 28
Neonatal : early neonatal mortality | from day 0 to day 6
Neonatal morbidity : immediate neonatal state | neonatal period
Neonatal morbidity : infection | neonatal period
Neonatal morbidity : respiratory disease | neonatal period
Neonatal morbidity : digestive disease | neonatal period

CONTACTS AND LOCATIONS:
Overall Officials: Gilles KAYEM, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Chenevier-Mondor, CHI, Créteil, France

REFERENCES:
- [Derived] Marcellin L, Batteux F, Chouzenoux S, Schmitz T, Lorthe E, Mehats C, Goffinet F, Kayem G. Second-trimester amniotic fluid proteins changes in subsequent spontaneous preterm birth. Acta Obstet Gynecol Scand. 2023 May;102(5):597-604. doi: 10.1111/aogs.14544. Epub 2023 Mar 14. PMID 36918342
- [Derived] Kayem G, Doloy A, Schmitz T, Chitrit Y, Bouhanna P, Carbonne B, Jouannic JM, Mandelbrot L, Benachi A, Azria E, Maillard F, Fenollar F, Poyart C, Bebear C, Goffinet F. Antibiotics for amniotic-fluid colonization by Ureaplasma and/or Mycoplasma spp. to prevent preterm birth: A randomized trial. PLoS One. 2018 Nov 7;13(11):e0206290. doi: 10.1371/journal.pone.0206290. eCollection 2018. PMID 30403730